CLINICAL TRIAL: NCT05565079
Title: Root Coverage Using Acellular Dermal Matrix and a Coronally Positioned Tunnel With or Without Biologic Materials
Brief Title: Root Coverage Using ADM and Coronally Positioned Tunnel With or Without Enamel Matrix Derivative
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Himabindu Dukka, Assistant Professor, DMD, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22.0637
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2024-04

CONDITIONS: Recession, Gingival
Keywords: esthetic surgery; allograft; biologic materials; acellular dermis
MeSH Terms: conditions — Gingival Recession | interventions — enamel matrix proteins

STUDY DESIGN:
Intervention Model Description: 24 patients will be recruited and randomly grouped as control or test treatment for root coverage using a coronally positioned flap and alloderm with (test) or without (control) enamel matrix derivative.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study involves an investigator (surgeon) and an examiner. The examiner measures the clinical parameters before and after surgery and is blinded to the surgical procedure and if the patient receives biologic materials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Coronally positioned tunnel with AlloDerm RTM and Enamel Matrix Derivative (Experimental): 12 patients will receive a coronally positioned tunnel with a regenerative tissue matrix (AlloDerm RTM, BioHorizons) and a porcine derived enamel matrix derivative (Emdogain, Straumann).
  Interventions: Biological: Regenerative tissue matrix and enamel matrix derivative; Biological: Regenerative tissue matrix
- Coronally positioned tunnel with AlloDerm RTM (Active Comparator): 12 patients will receive a coronally positioned tunnel with a regenerative tissue matrix (AlloDerm RTM, BioHorizons).
  Interventions: Biological: Regenerative tissue matrix

INTERVENTIONS:
Biological: Regenerative tissue matrix and enamel matrix derivative — Subjects in this group will receive a coronally positioned tunnel with a regenerative tissue matrix (AlloDerm, RTM) and a porcine-derived enamel matrix derivative (Emdogain).
  Other Names: Emdogain, Straumann
  Arms: Coronally positioned tunnel with AlloDerm RTM and Enamel Matrix Derivative
Biological: Regenerative tissue matrix — Subjects in both groups will receive a coronally positioned tunnel with a regenerative tissue matrix (AlloDerm, RTM).
  Other Names: AlloDerm RTM, BioHorizons

SUMMARY:
24 patients will be treated with a coronally positioned tunnel with AlloDerm RTM with or without the addition of Enamel Matrix Derivative to compare the baseline and 6-month changes in recession defect coverage, clinical attachment levels, amount of keratinized tissue width, and soft tissue thickness.

DETAILED DESCRIPTION:
Study Design: 24 patients will be treated: 12 with a coronally positioned tunnel with AlloDerm RTM (control), and 12 patients with a coronally positioned tunnel with Alloderm RTM and enamel matrix derivative (test). Included patients will undergo root coverage using the basic principles of a coronally positioned tunnel as described by Allen (2005). Six exams for measurements will be performed per patient: preoperative, two-week, one-, two-, four-, and six-months postoperatively.

Presurgical Management: Each patient will receive a diagnostic work-up, including standardized radiographs of the selected site and adjacent teeth (periapical and bitewing), clinical photographs, and a full mouth clinical examination. All women of childbearing potential will receive a pregnancy test. Presurgical preparation will include detailed oral hygiene instructions, scaling and root planing under local anesthesia, and occlusal adjustment (if indicated). Baseline data will be collected on the day of surgical treatment.

Clinical Measurements:

Baseline, two-week, one-, two-, four, and six-month data for the test site and adjacent dentition will include the following:

1. Miller's recession defect classification: Miller (1985).
2. Plaque index: Silness and Loe (1964).
3. Gingival index: Loe (1967).
4. Bleeding on probing index: Dichotomous scoring.
5. Gingival margin levels (Recession): Measured from CEJ to the gingival margin.
6. Keratinized tissue width: Measured from the gingival margin to the mucogingival junction.
7. Clinical attachment level: Measured from CEJ to the bottom of the clinical periodontal pocket.
8. Clinical tooth mobility: Modified Miller's Index, Laster (1975).
9. Radiographic examination: Paralleling technique with pre-operative periapical and bitewing radiographs.
10. Soft Tissue Thickness: Soft tissue measurements will be taken at three mid-buccal positions.
11. Tooth vitality: Tested with electric pulp tester and cold testing.
12. Patient models.
13. Clinical photographs.

Primary Outcome Variable 1. Site recession defect changes by comparing the pre- to the 6-month post-augmentation dimensions of soft tissues.

Secondary Outcome Variables

1. Site clinical attachment level changes by comparing the pre- to the 6-month post-augmentation sites.
2. Site gingival thickness changes by comparing the pre- to the 6-month post-augmentation dimensions of soft tissues.
3. Site keratinized tissue changes by comparing the pre- to the 6-month post-augmentation width of the keratinized soft tissues.

Surgical Treatment Treatment performed will be randomly assigned, via a coin toss, by the mentor at the beginning of the surgical appointment prior to local anesthesia. Root surfaces will be meticulously root planed using an ultrasonic instrument followed by hand instruments to obtain a smooth, hard root surface.

For control sites, the surgical procedure will consist of the preparation of a coronally positioned tunnel around the recession defect site without vertical releasing incisions. This technique is a modification of a previous tunnel technique described by Allen to include coronal positioning of the soft tissue over the allograft. The tissue will be elevated with a split-thickness incision beyond the mucogingival junction and extended until it is deemed enough release for tension-free coronal positioning of the tissue. The tunnel will be dissected with a microsurgical kit using loupes. The tunnel and AlloDerm RTM will extend one tooth mesial and distal to the recession site. Interproximal papillae will be elevated from the facial and lingual bone septum without papillary splitting incisions. The AlloDerm RTM will be positioned to completely cover the defect at the CEJ of the tooth and the inferior and lateral borders of the allograft will extend >3 mm beyond the osseous defect margins.

The test sites will be treated surgically in an identical manner for both tunnel preparation and AlloDerm graft placement. Additionally, enamel matrix derivative will be placed on the periosteal side of the soft tissue tunnel prior to placement and fixation of the ADM graft. Enamel matrix derivative will then be placed on both sides of the ADM prior to placement within the tunnel. After the graft and soft tissue have been secured in place, enamel matrix derivative will be placed over the entire area. For all sites, a monofilament polyglyconate Maxon 5-0 sling suture will be placed to maintain tensile strength for >6 weeks to secure the graft at the level of the CEJ. The marginal tissue will be placed as far coronal to the CEJ as possible to completely cover the AlloDerm graft and secured with sling sutures. Postoperative instructions will include: post-surgical regimen of at-home care instructions, 100 mg doxycycline hyclate qd for 14 days, 21 tablet 4 mg methylprednisolone dose pack, 600 mg ibuprofen q6h for 10 days, and 0.12% chlorhexidine gluconate bid for 10 days.

Surgical Measurements

1. Recession defect coverage (Initial recession depth, initial augmented, and post-augmented at 6 months):

   a. Direct= periodontal probe measurement from CEJ to gingival margin mid-defect.
2. Keratinized tissue height (Initial height, initial augmented, and post-augmented at 6 months)

   a. Direct= distance from the gingival margin to mucogingival junction stent. 16
3. Clinical attachment levels (Initial attachment loss and post-augmentation at 6 months)

   a. Direct= distance from the gingival margin to the base of periodontal pocket +/- distance from CEJ to the gingival margin.
4. Clinical photographs

Post-surgical patient management All patients will be seen at two weeks, one-, two-, four-, and six-months postoperative. Sutures will be removed between 4-8 weeks postoperatively. Postoperative visits will consist of supragingival plaque removal and oral hygiene reinforcement. Any patient who develops any significant post-operative complications, suffers an adverse reaction or allergy to the materials used, or shows attachment loss greater or > 2 mm on the treated tooth or adjacent teeth will be exited from the study and will receive appropriate treatment.

Potential risks:

There are known physical risks linked with root coverage procedures and the placement of soft tissue allografts. These risks include:

1. Infection of the treated area
2. Mild bruising and/or bleeding
3. Mild swelling
4. Transient or, rarely, permanent tooth sensitivity to hot, cold, sweet, or acidic foods
5. Transient or, rarely, permanent paresthesia or numbness of lips, tongue, chin, or gums
6. Loss of the soft tissue graft with occasionally more recession or increased spacing between teeth
7. Allergic reaction to the soft tissue graft
8. Accidental swallowing of foreign matter

There may also be additional, unforeseen risks involved with these procedures. In terms of economic risk, if the treatment fails, the patient will be retreated at no charge in the Graduate periodontics clinic. In terms of legal risks, if the patient is injured as a result of his/her participation in this study, treatment for the injury will be provided at the University of Louisville Hospital. The patient or the patient's insurance company will be billed for the costs of such medical treatment. Additional compensation, for things such as lost wages, inconvenience, or discomfort will not be provided.

Adverse events:

1. An "adverse event" refers to any adverse experience occurring during the clinical study period, whether associated or not associated with the study test articles or procedures.
2. A "serious adverse event" means any experience that suggests a significant hazard, contraindication, side effect, or precaution. With respect to human clinical experience, a serious adverse event includes any experience that is fatal or life-threatening, causes a persistent or permanent disability, requires initial or prolonged hospitalization, requires medical or surgical intervention to prevent permanent impairment or damage, or is a congenital anomaly.
3. An "unanticipated adverse event" is one that is not identified in nature, severity, or frequency in the investigator's brochure.

Adverse events will be collected by observing and interviewing the subject during the study. Subjects who experience any significant problems during the study are to call and discuss them with the investigator. Any suspected adverse event or allergic response is to be thoroughly examined by the investigator. All adverse events are to be reported. All subjects experiencing adverse events will be followed by the investigator until there is a return to the subject's baseline condition or a clinical satisfactory resolution is achieved.

Adverse events which are serious or unanticipated are to be reported immediately by phone to the study director and promptly reported to IRB (within five working days of the UofL site awareness) through completion of the Serious Adverse Event (SAE) Reporting Form within the ESS system, which includes the date of the event, description of the adverse event, involved study treatment, and outcome of the event. Examples of expected, but rarely occurring adverse events related to grafting treatment include clinical observation of infection, flap necrosis, severe inflammation, and severe pain. Additionally, unanticipated problems (UPIRTSOs) require completion of teh UPIRTSO Reporting Form within the ESS system to IRB.

If the IRB requests any additional data or information regarding the reported events, Follow-Up Reports and Response to Stipulations will be reported within 15 working days after receiving the IRB request.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one Miller class 1 or 2 soft tissue recession defect >3 mm on a non-molar tooth.
* Healthy patients, at least 18 years of age.
* Patient understands and signs an informed consent approved by the University of Louisville IRB.

Exclusion Criteria:

* Patients with debilitating systemic diseases, diseases that significantly affect the periodontium, infectious diseases, or psychological problems that may interfere with treatment.
* Previous head and neck radiation or chemotherapy within the previous 12 months.
* Patients with known allergies to any of the materials used in the study, including systemic antibiotics.
* Patients that use tobacco products (smoking, smokeless tobacco, or electronic cigarettes).
* Patients with alcohol abuse problems.
* Patients requiring antibiotic prophylaxis for dental procedures.
* Cemento-enamel unction not identifiable.
* Root surface restorations at the recession site.
* Patients undergoing long-term steroid therapy.
* History of previous root coverage procedure, graft, or guided tissue regeneration involving the recession site.
* Pregnant or lactating patients.
* Patients who fail to maintain oral hygiene levels of at least 80% plaque-free surfaces.
* Patients who fail to complete the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Recession defect coverage | 6 months
  To compare baseline and 6-month changes in recession defect coverage

SECONDARY OUTCOMES:
Clinical attachment levels | 6 months
  To compare baseline and 6-month changes in clinical attachment levels
Keratinized tissue width | 6 months
  To compare baseline and 6-month changes in amount of keratinized tissue
Soft tissue thickness | 6 months
  To compare baseline and 6-month changes in soft tissue thickness

CONTACTS AND LOCATIONS:
Overall Officials: Bindu Dukka, BDS, MSD, MPH, Principal Investigator — Director, Graduate Periodontics, University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aroca S, Keglevich T, Nikolidakis D, Gera I, Nagy K, Azzi R, Etienne D. Treatment of class III multiple gingival recessions: a randomized-clinical trial. J Clin Periodontol. 2010 Jan;37(1):88-97. doi: 10.1111/j.1600-051X.2009.01492.x. Epub 2009 Nov 30. PMID 19968743
- [Result] Vincent-Bugnas S, Charbit Y, Lamure J, Mahler P, Dard MM. Modified Tunnel Technique Combined with Enamel Matrix Derivative: A Minimally Invasive Treatment for Single or Multiple Class I Recession Defects. J Esthet Restor Dent. 2015 May-Jun;27(3):145-54. doi: 10.1111/jerd.12170. PMID 26094684
- [Result] Shepherd N, Greenwell H, Hill M, Vidal R, Scheetz JP. Root coverage using acellular dermal matrix and comparing a coronally positioned tunnel with and without platelet-rich plasma: a pilot study in humans. J Periodontol. 2009 Mar;80(3):397-404. doi: 10.1902/jop.2009.080438. PMID 19254123